CLINICAL TRIAL: NCT03134651
Title: The Effect of Preoperative Anxiety With Depth of Anesthesia During Oocyte Retrieval on IVF Success
Brief Title: Preoperative Anxiety at Oocyte Retrieval
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Sevtap Hekimoglu Sahin, Clinical Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUTF-GOKAEK 2014/115
Record Dates: First submitted 2017-03-30; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Infertility, Female; Anesthesia Awareness; Anxiety State
Keywords: Anxiety; Oocyte retrieval; Monitoring of brain function
MeSH Terms: conditions — Infertility, Female; Intraoperative Awareness; Anxiety Disorders | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monitoring brain function-low-anxiety (Active Comparator): Anxiety has determined a cutoff score of 17. Patients were divided into two groups according to the recorded BAI score: a low-anxiety group and a high-anxiety group.The monitoring brain function values were recorded at baseline, 5 minutes, 15 minutes, and after anesthesia. Propofol was performed by ventilation with face mask. Monitoring brain function was keep value between 40 and 60.
  Interventions: Device: Monitoring brain function; Drug: propofol
- monitoring brain function-high-anxiety (Active Comparator): Anxiety has determined a cutoff score of 17. Patients were divided into two groups according to the recorded BAI score: a low-anxiety group and a high-anxiety group.The monitoring brain function values were recorded at baseline, 5 minutes, 15 minutes, and after anesthesia. Propofol was performed by ventilation with face mask. Monitoring brain function was keep value between 40 and 60.
  Interventions: Device: Monitoring brain function; Drug: propofol

INTERVENTIONS:
Device: Monitoring brain function
Drug: propofol
  Other Names: propofol %1

SUMMARY:
This study evaluated the effects of preoperative anxiety and dosage of anesthesia on IVF success. Half of participants according to the recorded Beck's Anxiety Inventory (BAI) score: a low-anxiety group, while the other half high-anxiety group.

DETAILED DESCRIPTION:
Anxiety is common among women hospitalized for oocyte retrieval. Infertility is usually accompanied by psychological and behavioral changes and can result in preoperative anxiety. Sometimes, preoperative anxiety can be serious. Furthermore, in the absence of premedication for oocyte retrieval, severe degrees of anxiety may occur. Anxiety effects the total consumption of analgesic and anesthetic drugs intraoperatively and has a negative impact on recovery from anesthesia. In addition, the negative effect of anesthetic agents used on fertilization and embryo quality during in vitro fertilization (IVF) has been discussed. However, the impact of any of them on fertilization and embryo quality has not been clearly determined to date. Studies have reported different results regarding the negative effects of anesthetic agents on embryo development and fertilization.

ELIGIBILITY:
Inclusion Criteria:

* oocyte retrieval under sedation
* 25 and 43 years of age
* American Society of Anesthesiologists physical status I-II

Exclusion Criteria:

* history of psychiatric illness
* secondary infertility can be surgically corrected
* not able to communicate well in the native language
* those women who necessitated general anesthesia

Ages: 25 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — infertile women
Enrollment: 131 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2016-07-24 (Actual); Study Completion 2016-09-24 (Actual)

PRIMARY OUTCOMES:
Changes in perioperative Monitoring brain function were measured | Preoperative, intraoperative and postoperative first minute
  Monitoring brain function was assessed Change from baseline at preoperatively, intraoperative 5th and 15th minutes and after anesthesia

SECONDARY OUTCOMES:
pregnancy rate | 10 days
  pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: Sevtap Hekimoglu Sahin, Professor, Study Chair — Trakya University Medical Faculty

IPD SHARING:
Plan to Share IPD: No